CLINICAL TRIAL: NCT06596824
Title: Personalized Digital Training Intervention to Reduce Inflammation by Correcting Pathological Movement Patterns in Pre-stage Knee Osteoarthritis (OA)
Brief Title: Personalized Digital Training Intervention to Reduce Inflammation by Correcting Pathological Movement Patterns in Pre-stage Knee Osteoarthritis After Anterior Cruciate Ligament Reconstruction
Acronym: PROTO-WP4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Tobias Winkler, Prof. Dr.med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROTO-WP4; 101095635 (Other Grant/Funding Number: Horizon-Programm der EU)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis (OA) of the Knee; ACL Reconstruction
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The treatment group (Experimental): In addition to the standard-of-care physiotherapy program, the treatment group will additionally receive a training intervention utilizing sensor-based technology that provides 3D avatar training, supported by an accompanying app, to deliver personalized exercise regimens. This intervention aims to correct the pathological knee movement and loading patterns that exacerbate joint inflammation and contribute to the development of knee OA.
  Interventions: Behavioral: Training intervention
- the control group (No Intervention): Standard-of-care physiotherapy program

INTERVENTIONS:
Behavioral: Training intervention — Personalized digital training intervention aims to correct pathological knee movement and loading patterns and reduce inflammation in pre-stage knee osteoarthritis.
  Arms: The treatment group

SUMMARY:
Osteoarthritis (OA) is a condition that causes pain and stiffness in the joints, often due to injuries like torn ligaments. Even after surgery, these injuries can lead to long-term joint problems. Current treatments don't fully prevent OA from developing. This study is testing a new 12-week exercise program designed to improve how the knee moves, using a special sensor-based system. The goal is to reduce joint inflammation and prevent the development of OA in patients who have had knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Underwent anterior cruciate ligament reconstruction (ACLR) due to an acute knee injury in the past 12 months
* ACLR patients with aberrant gait profiles who exhibit all three aberrant characteristics (knee flexion angle, knee flexion moment, and knee adduction moment)

Exclusion Criteria:

* Previous trauma or surgery (other than ACLR) to any weight-bearing joint,
* Signs of knee OA as defined by the OARSI-Joint Space Narrowing (JSN) Score of two or more (standing AP x-ray)
* Body mass index ≥ 30 kg/m2;
* Inflammatory arthropathies;
* Immunosuppression due to illness or medication;
* Sepsis or hemostasis disorders;
* Severe uncontrolled inflammatory disease or autoimmune disease (e.g., ulcerative colitis, Crohn's disease, etc.);
* Having malignancy and undergoing treatment including chemotherapy, radiotherapy, or immunotherapy;
* Unable to freely give their informed consent (e.g., individuals under legal guardianship).
* Currently enrolled in or has not yet completed a period of at least 5 times as the half-life time of the drug used in the previous trial since ending other investigational device or drug trial(s)
* Patients who are dependent on the sponsor, investigator, or study site;
* Pregnant or breast-feeding women or women of childbearing potential not protected by an effective contraceptive method of birth control (defined as pearl index < 1);
* Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel;
* Patients who are committed to an institution by virtue of an order issued by either the judicial or the administrative authorities;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | at 6-month follow-up visit
  Restoration of normal knee angle and moment patterns during walking at 6-month follow-up (compared to normative data), as determined by a machine learning-derived gait index.

SECONDARY OUTCOMES:
Secondary endpoints measure the potential magnetic resonance imaging (MRI) changes from BL for the following parameters: | Baseline, 6, and 36 months followup visits
  MRI parameters are chosen to assess the potential patient response as an indicator of intervention efficacy. The aim is to examine the longitudinal association between knee biomechanics parameters and MRI-based measures of inflammation/degradation. The following MRI parameters will be checked:
  * Quantitative composition of cartilage
  * Quantitative morphology of the cartilage
  * The degree of synovitis and effusion
  * Semi-quantitative measurements of structural pathology (MRI Osteoarthritis Knee Score)

OTHER OUTCOMES:
Exploratory Endpoints measure the potential changes from BL for the following parameters: | Baseline, 6, and 36 months follow-up visits
  Cellular and molecular biomarker profiling defines patients' BL biomarker profiles and identifies any potential difference after the intervention. The aim is to examine the longitudinal association between knee biomechanics parameters and the possible change in the following parameters.
  * Biomarker analysis in blood and urine specimens
  * Biomarker analysis in synovial fluid (SF) specimens

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No